CLINICAL TRIAL: NCT04090775
Title: A Phase 2 Trial of Cryosurgical Freezing and Intratumoral Combination Immunotherapy in Men With Metastatic Prostatic Adenocarcinoma
Brief Title: A Phase 2 Trial for Men With Metastatic Prostatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rampart Health, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSCOPAL 1001
Record Dates: First submitted 2019-08-09; First posted 2019-09-16 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-02

CONDITIONS: Metastatic Prostatic Adenocarcinoma
MeSH Terms: interventions — Nivolumab; Ipilimumab; Cyclophosphamide; Cryosurgery

STUDY DESIGN:
Intervention Model Description: Male subjects greater than 18 years of age with histologically-proven cancer of the prostate with at least one imaging- or histologically -proven metastasis to lymph nodes or bone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm. Subjects receiving treatment. (Other): Cryosurgical freezing and intratumoral combination immunotherapy as determined by the proportion of patients achieving serum PSA decline from baseline of at least 50%.
  Interventions: Drug: Opdivo Injectable Product; Drug: Yervoy Injectable Product; Drug: Cytoxan; Procedure: Cryosurgical freezing (cryosurgery)

INTERVENTIONS:
Drug: Opdivo Injectable Product — Opdivo (nivolumab): PD-1 inhibitor antibody
  Injectable 10mg/mL, only 1 mL injected.
  Other Names: nivolumab
Drug: Yervoy Injectable Product — Yervoy (ipilimumab): Anti-CTLA-4 antibody
  Injectable 5mg/mL, only 1 mL injected.
  Other Names: ipilimumab
Drug: Cytoxan — Cytoxan (cyclophosphamide): Chemotherapy agent
  Both Injectable and Oral low dose:
  Injectable 250mg/m2, only 1 mL injected. Oral low dose cyclophosphamide: option of either 50mg once daily pill or 25mg twice daily pill for two weeks on, then two weeks off, then two weeks on again.
  Other Names: Cyclophosphamide
Procedure: Cryosurgical freezing (cryosurgery) — Cryosurgery, also known as cryoablation, for prostate cancer works by freezing the cancer cells inside the prostate gland. Cryoablation will release intact antigens to prime the immune system.
  Other Names: Cryoablation

SUMMARY:
This study seeks to estimate the occurrence of adverse events related to the study treatment (Cryosurgical freezing and Intratumoral Combination Immunotherapy), as well as determine the potential efficacy.

DETAILED DESCRIPTION:
Cryosurgical freezing will release intact antigens to prime the immune system. The study treatment immunotherapeutic drugs (PD-1 inhibitor monoclonal antibody nivolumab and anti-CTLA-4 monoclonal antibody ipilimumab, and cyclophosphamide) will then be sequentially injected directly into the cancer immediately following cryosurgical freezing. Oral low-dose cyclophosphamide will also be administered subsequently. It is speculated that neoantigens released from the cryoablated necrotic cancer will be available in the vicinity of the cryosurgical freezing field immediately following the procedure. Immature dendritic cells attracted to the injection site will internalize neoantigens to become activated to recognize cancer-specific antigenic proteins. The activated dendritic cells will recruit killer T-cells to the injection site to attack cancer cells, and then migrate through the lymphatic system to sites of metastases, targeting cancer-specific neoantigens and recruiting more killer T-lymphocytes to destroy other cancer cells harboring the precise antigenic epitopes (abscopal (bystander) effect). In this way, dendritic cells are capable of initiating cell-mediated systemic immune response in combination with cytotoxic killer T-cells. Regulatory T lymphocytes, which have been implicated in dampening or halting cell-mediated, antigen-specific immune responses, will be selectively depleted by anti-CTLA-4 monoclonal antibodies and low-dose cyclophosphamide. Intratumoral injection of the immunotherapeutic medications assists in stimulating and harnessing the local and systemic immune response. Oral cyclophosphamide prolongs the immune response. Using this combination of therapies, referred to as AbscopalRx1001, it is thought that a clinically significant systemic anti-cancer immune response might be elicited. Intratumoral injection of drugs will likely offer fewer side effects than systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

5.3.1 Be willing and able to provide written informed consent/assent for the trial.

5.3.2 Be ≥18 years of age on day of signing informed consent.

5.3.3 Have a performance status of 0-3 on the ECOG Performance Scale.

5.3.4 Have a life expectancy of 6 months or more as determined by treating physician.

5.3.5 Not a candidate for or refuses chemotherapy; or failure of prior chemotherapy.

5.3.6 PSA >2 ng/mL at baseline.

5.3.7 Available archival tumor tissue for correlative studies. Submission of archival TRUS prostate biopsy tissue is required if available, in the form of representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (preferred) or at least 15 slides, with an associated pathology report. If archival prostate tissues are unavailable or cannot be obtained, a repeat TRUS prostate biopsy is not required for eligibility.

5.3.8 Histologically-documented adenocarcinoma or mixed adenocarcinoma-neuroendocrine carcinoma of the prostate. All subjects must submit their primary tumor or metastatic biopsy pathology specimens and laboratory and imaging reports to Rampart Health where they will be centrally reviewed. Central Rampart Health pathologic review is not required for screening but rather for confirmation of diagnosis and histologic subtype of cancer. Local pathologic review is sufficient for eligibility determination.

5.3.9 Measurable disease as defined by PCWG3 using iRECIST criteria and identified by radiographic imaging. In order to be eligible, the patient must have at least one metastatic bone and/or metastatic lymph node site(s) with cancer mass measuring 1 cm or more in diameter based on bone and/or soft tissue lesions as defined by any of the following:

* Bone metastases defined by bone imaging. If the patient has technetium bone scan, and/or NaF PET performed, either study may be used for documenting metastases; both scans do not need to show the number of metastases required for study entry. For patients undergoing PSMA PET, only PSMA avid lesions that are consistent with metastasis will be counted as a site of metastasis.
* Distant metastatic lymph node disease defined by imaging. A lymph node ≥1 cm in shortest dimension will be noted as involved with disease. Distant metastatic lymph nodes will be determined as any lymph nodes outside the confines of the true pelvis. For patients undergoing PSMA PET, only PSMA avid lesions that are consistent with metastasis will be counted as a site of metastasis.
* Any other soft tissue lesion defined by imaging deemed by the physician to be consistent with distant metastatic disease. For patients undergoing PSMA PET, only PSMA avid lesions that have a CT or MRI correlate consistent with metastasis will be counted as a site of metastasis.

5.3.10 The effects of the medications in this protocol on the developing human fetus are unknown. Men treated or enrolled on this protocol must agree to use adequate contraception prior to the first dose of study therapy, for the duration of the study participation, and for 120 days after the last dose of study therapy.

5.3.11 Their partners should be encouraged to use proper method of contraception.

5.3.12 Acceptable initial laboratory values within 14 days of treatment initiation according to the following: ANC ≥ 1500/µl; Hemoglobin ≥ 9.0 g/dL(prior transfusion permitted); Platelet count ≥ 100,000/µl; Creatinine ≤ 2.0 x the institutional upper limit of normal (ULN) OR creatinine clearance >30 ml/min; Potassium ≥ 3.5 mmol/L (within institutional normal range); Bilirubin ≤ 1.5 x ULN (unless documented Gilbert's disease); SGOT (AST) ≤ 2.5x ULN, or <5x ULN in patients with documented liver metastases; SGPT (ALT) ≤ 2.5x ULN or <5x ULN in patients with documented liver metastases; Albumin >2.5 mg/dL; Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. Deviation from these values is allowed at the discretion of the treating investigator.

5.3.13 No active major medical or psychological problems that could be complicated by study participation.

Exclusion Criteria:

5.4.1 Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.

5.4.2 Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment, with the exception of steroids for adrenal insufficiency in which case prednisone <10mg/day or its equivalent is allowed.

5.4.3 Has a performance status of 4-5 on the ECOG Performance Scale.

5.4.4 Has a known history of active TB (Bacillus Tuberculosis).

5.4.5 Hypersensitivity to monoclonal antibodies such as nivolumab or any of its excipients.

5.4.6 Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.

5.4.7 Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.

5.4.8 Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Persisting toxicity related to prior therapy (NCI CTCAE v.5 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, Grade 2 anemia, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.

5.4.9 Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting.

5.4.10 Has a known additional malignancy that is progressing or requires active treatment. Exceptions include carcinoid, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

5.4.11 Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs), including but not limited to systemic or cutaneous lupus erythematosus, cutaneous psoriasis, psoriatic arthritis, rheumatoid arthritis, scleroderma, sicca syndrome, polymyalgia rheumatica, polyarteritis nodosa, granulomatous polyangiitis, microscopic polyangiitis, polyarteritis nodosa, temporal arteritis, giant cell arteritis, dermatomyositis, Kawasaki disease. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, hydroxychloroquine, etc.) is not considered a form of systemic treatment.

5.4.12 Has known history of, or any evidence of active, non-infectious pneumonitis.

5.4.13 Has an active infection requiring systemic therapy.

5.4.14 Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

5.4.15 Has known psychiatric or substance abuse disorder or any other condition that would interfere with cooperation with the requirements of the trial in the opinion of the Physician-investigator.

5.4.16 Expecting to father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

5.4.17 Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

5.4.18 Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

5.4.19 Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed within 30 days.

5.4.20 Personal representative (family member or friend) withholds consent for any reason.

5.4.21 Unable for any reason to understand the consent form and other written information and freely give written informed consent.

5.4.22 Scores less than 14.5 (out of possible maximum of 20) on the UBACC Capacity to Consent Assessment Instrument.

5.4.23 Does not re-sign the consent form a second time at least 24 hours after initial consent but before the treatment procedure.

5.4.24 Hypersensitivity to Cyclophosphamide.

5.4.25 Urinary outflow obstruction.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: PSA decline | baseline to 8 weeks after end of treatment (approximately 6 months)
  Primary Endpoint: Efficacy of cryosurgical freezing and intratumoral combination immunotherapy as determined by the proportion of patients achieving serum PSA decline from baseline of at least 50%.

SECONDARY OUTCOMES:
Efficacy of cryosurgical freezing and intratumoral combination immunotherapy iRECIST criteria | baseline to 8 weeks after end of treatment (approximately 6 months)
  Efficacy of cryosurgical freezing and intratumoral combination immunotherapy as determined by iRECIST criteria. Overall response rate as determined by PCWG3 using iRECIST radiographic response.

OTHER OUTCOMES:
Efficacy of cryosurgical freezing and intratumoral combination immunotherapy RECIST 1.1 Criteria | baseline to 8 weeks after end of treatment (approximately 6 months); quarterly up to one year; and thereafter biannually for up to 2 more years.
  Efficacy of cryosurgical freezing and intratumoral combination immunotherapy as determined by RECIST1.1 criteria. Overall response rate as determined by PCWG3 using RECIST1.1 radiographic response.
Radiographic progression-free survival (rPFS) | baseline to 8 weeks after end of treatment (approximately 6 months); quarterly up to one year; and thereafter biannually for up to 2 more years.
  Radiographic progression-free survival (rPFS) rPFS as determined by PCWG3 with both RECISTS1.1 and iRECIST criteria.
Best overall response of confirmed PR or CR by independent radiology review | From signing of Informed Consent form, approximately every 4 weeks for the first 3 months; quarterly up to one year; and thereafter biannually for up to 2 more years.
  Best overall response of confirmed PR or CR by independent radiology review
Time to Prostate Specific Antigen (PSA) progression (TTPP) | Baseline up to 8 weeks after last treatment; quarterly up to one year; and thereafter annually for up to 2 more years.
  Time to Prostate Specific Antigen (PSA) progression (TTPP) Time to PSA progression is measured from the date of first study treatment until the date of PSA progression according to PCWG3 criteria.
Overall survival | 3 years
  Overall survival: Number and percent of participants that are alive.
Incidence of AEs/SAEs | baseline to 8 weeks after the last treatment; quarterly up to one year; and thereafter biannually for up to 2 more years.
  Incidence of AEs/SAEs: An AE is any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity. Incidence was defined as the number of participants who experienced an adverse event within their period of participation in this study. Incidence of adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Severity of AEs/SAEs | baseline through 8 weeks after the last treatment; quarterly up to one year; and thereafter biannually for up to 2 more years.
  Severity of AEs/SAEs
Duration of AEs/SAEs | baseline through 8 weeks after the last treatment; quarterly up to one year; and thereafter biannually for up to 2 more years.
  Duration of AEs/SAEs

CONTACTS AND LOCATIONS:
Overall Officials: David G Bostwick, M.D.,M.B.A., Principal Investigator — Rampart Health
Locations (2):
- United States (2):
  - Antelope Valley Urology & Incontinence, Lancaster, California
  - Ascension Providence Rochester Hospital, Rochester, Michigan